CLINICAL TRIAL: NCT06700785
Title: A Pharmacokinetic Comparison of Three Butyrate Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BUTY-0324-01
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — lysine butyrate; Butyric Acid; tributyrin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lysine Butyrate (Experimental)
  Interventions: Dietary Supplement: Lysine butyrate
- Sodium buytrate (Active Comparator)
  Interventions: Dietary Supplement: Sodium Butyrate
- Tributyrin (Active Comparator)
  Interventions: Dietary Supplement: Tributyrin

INTERVENTIONS:
Dietary Supplement: Lysine butyrate — Lysine butyrate supplement. This study will compare plasma pharmacokinetic profiles of three commercially available butyrate supplements.
  Arms: Lysine Butyrate
Dietary Supplement: Sodium Butyrate — Oral sodium butyrate supplement.
  Arms: Sodium buytrate
Dietary Supplement: Tributyrin — Oral tributyrin supplement.
  Arms: Tributyrin

SUMMARY:
This study is a randomized, three-arm, interventional study of N=10 apparently healthy men. This study will quantify plasma butyrate responses to a single dose of three different butyrate products.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 25 and 45 (inclusive).
* Body Mass Index of 18.5-24.9 (inclusive).
* Body weight of at least 110 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5-minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from alcohol, caffeine, and exercise for 24 hours and fast for 10 hours prior to each of the treatments.
* Participant agrees to maintain existing dietary and physical activity patterns throughout the study period.
* Participant is willing and able to comply with the study protocol.

Exclusion Criteria:

* A history of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal disease.
* The participant's alcohol consumption is more than two standard alcoholic drinks per day or more than 10 drinks per week or has a history of drug/alcohol abuse or dependence.
* History of diabetes (any form) or any endocrine disorder.
* Fasting blood sugar of > 125 mg/dL.
* Current smokers or smoking cessation within the past month (28 days).
* History of hyperparathyroidism or an untreated thyroid disease.
* History of malignancy in the previous five years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Any history of gastrointestinal bypass surgery, etc., or any known functional gastrointestinal disorder that may impact nutrient absorption, e.g., short bowel syndrome, atrophic gastritis, IBD, diarrheal illnesses, history of colon resection, gastroparesis, gastric resection, celiac disease, or Inherited Errors of Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g., rheumatoid arthritis, Crohn's Disease, ulcerative colitis, lupus, HIV/AIDS, etc.).
* History of using butyrate or tributyrin-containing dietary supplements within the past seven days.
* Known allergy or sensitivity to any ingredient in the test formulations as listed on the product label.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
plasma butyrate levels | Prior to product administration (time 0), as well as 20, 45, 90, 150, and 210 minutes post-dose
  Plasma butyrate levels in ug/mL.

SECONDARY OUTCOMES:
Visual analog scales for cognitive function. | 0, 20, 45, 90, 150 and 210 minutes post-dose
  Cognitive function as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better cognitive function.
Visual analog scales for mood. | 0, 20, 45, 90, 150 and 210 minutes post-dose
  Mood as measured by a traditional 10 cm visual analogue scale (VAS), where values can range from 0 to 10, and higher values represent better mood.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided